CLINICAL TRIAL: NCT04200183
Title: iACT With Pain: an ICT-delivered Intervention for Self-management of Chronic Pain
Acronym: iACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Paula Castilho, Assistant Professor, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTDC/PSI-GER/28829/2017
Record Dates: First submitted 2019-09-18; First posted 2019-12-16 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Chronic Pain
Keywords: chronic pain; contextual behavioral intervention; acceptance and commitment therapy; mindfulness; compassion-based therapy; online intervention
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iACTwithPain (Experimental)
  Interventions: Behavioral: iACTwithPain (ACT+compassion)
- ACT-only intervention (Experimental)
  Interventions: Behavioral: ACT-only intervention
- Wait list (inactive control) (No Intervention)

INTERVENTIONS:
Behavioral: iACTwithPain (ACT+compassion) — This intervention will deliver a eHealth ACT and compassion-based therapy (iACTwithPain) designed for chronic pain
  Arms: iACTwithPain
Behavioral: ACT-only intervention — This intervention will deliver the iACTwithPain intervention but without the delivery of explicit compassion.
  Arms: ACT-only intervention

SUMMARY:
This project aims to test the effectiveness of an ICT-based delivery of an evidencebased psychological intervention for Chronic Pain (CP) - iACTwithPain. CP is a prevalent health problem worldwide, including in Portugal (around 30% of population) placing a significant economic burden on healthcare systems. Although CP is associated with psychological symptoms (i.e. depression and anxiety) and poor social functioning and quality of life, there is a lack of nationwide provision of evidence-based psychological services in healthcare units for CP. Information and Communication Technologies (ICTs) offer attractive tools through which self-management programmes can be delivered. The dissemination and commercialization of iACTwithPain will provide a much-needed pain self-management service and its ICT-based delivery form will increase the accessibility in large cohorts of the population with limited access to standard treatment.

DETAILED DESCRIPTION:
This project aims to develop and deliver an ICT self-management intervention for chronic pain (CP)-iACT. As persistent pain of different etiologies represents a medical, social and economic burden, optimized management of pain tools to support CP patients in adjusting to their condition and improving quality of life is timely and can lead to more costeffective healthcare systems by promoting the management of CP outside health institutions.

While CP influences and is influenced by psychological factors, provision of care to CP patients in Portugal vastly disregards psychological interventions. In contrast, the usual treatment to CP in Portugal is primarily pharmacologic, which has limited effects. Psychological interventions are well suited for addressing the cognitive, emotional and behavioral factors that contribute to and result from pain-related distress. Acceptance and Commitment Therapy(ACT) is an evidence-based psychological approach for CP. ACT focuses on fostering acceptance of the unavoidable aspects of pain and directing efforts towards behavioral functioning, rather than the traditional focus on controlling pain, which disregards the patient's overall functioning and well-being.

Also, studies suggest that self-compassion mediate the change in disability and psychopathological symptoms in ACT interventions for CP, although self-compassion is not a specific target in ACT. Thus, an explicit focus on self-compassion might increase the efficacy of ACT interventions, although this hypothesis has not been tested.

Online interventions have several advantages: reducing therapist time and waiting lists, increased cost-effectiveness, patients working at their own pace, accessibility to large clinical samples and rural and remote clinical cohorts.

However, evidence for the effectiveness of online-delivered ACT for CP is still scarce, with only three studies with several methodological limitations (i.e. small sample size and non-randomization). The innovative features of the current project are:1)the development of an ICT solution for self-management of pain, and improvement of overall well-being tailored to CP patients;2) the improvement of an ACT intervention by including psychological symptoms, and the increase in overall functioning and quality of life of CP patients; b)adding a new component(self-compassion) to the intervention will increase its effectiveness;c) its format will be a cost-effective solution for self-management of CP. The research strategy to achieve the project's goals follows a randomized controlled trial design with three arms: 1.iACTwithPain intervention (ACT + self-compassion); 2. ACT-only intervention; 3.Waiting List. iACTwithPain may also impact on other spheres of patients' lives such as work (e.g.,less absenteeism) and social (e.g.,less restrictions for leisure activities), which will contribute to more social inclusion.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 50;
* a CP diagnosis at least for the last three months;
* access to internet and willingness to do it regularly (at least once a week)
* willingness to be randomized
* provide informed consent.

Exclusion Criteria:

* undergoing any other form of psychological intervention for CP;
* severe psychiatric problem (e.g. severe depression; psychotic illness; bipolar disorder; borderline personality disorder), assessed using several questions (self-reported) based on the diagnostic criteria according to DSM-V;
* pain due to malignancy, trauma, or surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 246 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain impact. | baseline, 8 weeks, 3 months, 6 months
  The 6-item Pain Impact Questionnaire (PIQ-6 (52,53) ) will be used to assess participants' perceived pain severity (1 item rated on a 6-point scale) and impact on emotional well-being, leisure activities, and work functioning (5 items rated on a 5-point scale).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carvalho SA, Trindade IA, Duarte J, Menezes P, Patrao B, Nogueira MR, Guiomar R, Lapa T, Pinto-Gouveia J, Castilho P. Efficacy of an ACT and Compassion-Based eHealth Program for Self-Management of Chronic Pain (iACTwithPain): Study Protocol for a Randomized Controlled Trial. Front Psychol. 2021 Mar 9;12:630766. doi: 10.3389/fpsyg.2021.630766. eCollection 2021. PMID 33767648